CLINICAL TRIAL: NCT07268716
Title: A Randomized Controlled Clinical Trial to Assess the Efficacy of Tailored Patient Information and Voluntary Patient-Managed Outpatient Digital Follow-Up as an Adjunct to Standard Treatment According to National Guidelines in Adult Trauma Patients in Norway (The POSTRAUMA Trial).
Brief Title: Assess the Efficacy of Tailored Patient Information and Voluntary Patient-managed Outpatient Digital Follow-up (I-POD) as an Adjunct to Standard Treatment According to National Guidelines in the National Trauma Plan Among Adult Trauma Patients in Norway.
Acronym: POSTRAUMA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 909877
Record Dates: First submitted 2025-11-25; First posted 2025-12-08 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-11

CONDITIONS: Trauma Centers; Trauma Patients; Trauma (Including Fractures); Trauma Injury; Rehabilitation After Neurological or Orthopaedic Injuries; Rehabilitation; Return to Work; HRQOL (Health Related Quality Of Life); EQ5D5L-VAS
Keywords: multitrauma; trauma; rehabilitation; return to work; HRQOL; EQ5D
MeSH Terms: conditions — Wounds and Injuries; Accidental Injuries

STUDY DESIGN:
Intervention Model Description: Randomized controlled clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Standard treatment and follow up after trauma according to national guidelines in the National trauma plan.
- Intervention group (Active Comparator): Tailored patient information and patient-managed outpatient follow up as an adjunct to standard treatment according to national guidelines in the National trauma plan
  Interventions: Other: The intervention is a tailored patient Information and Patient-managed Outpatient Digital follow-up treatment

INTERVENTIONS:
Other: The intervention is a tailored patient Information and Patient-managed Outpatient Digital follow-up treatment — The objective of the POSTRAUMA-trial is to assess if the I-POD intervention combined with standard treatment according to national guidelines, lead to less disability measured by EQ5D-index, better health-related quality of life measured by EQ-VAS and increased return to studies and work compared to standard treatment after trauma.
  Other Names: I-POD intervention
  Arms: Intervention group

SUMMARY:
The POSTRAUMA trial is a clinical trial at The Regional trauma centre of Western Norway, Haukeland University Hospital.

Trauma is the leading cause of death worldwide in patients aged 1-45 years. In Norway, approximately 10,000 patients are admitted to hospital annually due to trauma, with 66% being male. The mean age is 43 years for male and 48 years for female, indicating a relatively young patient population.

While mortality rates are decreasing, a significant proportion of trauma survivors experience long-term disabilities, reduced quality of life, and difficulties in returning to work. These consequences impose substantial burdens on individuals, families, and society. Considering these issues, a shift in focus is needed-from survival alone to long-term functional recovery and quality of life after trauma.

Severe trauma often requires long-term follow-up, both physically and psychosocially. Traditional follow-up can be fragmented and not tailored to individual needs. Digital patient monitoring and tailored information have the potential to improve patient pathways, but knowledge about how these are experienced by patients is limited.

The goal is to find out if Norwegian trauma patients who receive tailored patient information and patient-managed outpatient digital follow-up, in addition to standard treatment have:

* Less disability
* Return more often to work
* Improved quality of life

The study population are Norwegian trauma patients, 16 years or older at date of inclusion, who are admitted to Haukeland University hospital (HUS) following trauma with trauma team activation. 256 patients will be included in this trial.

Participants will:

* Answer a questionnaire at inclusion, one month, 6 months and 12 months.
* Participants in the intervention group will be invited to digital outpatient follow up one month after the accident.
* Some participants will be interviewed about how they experienced their trauma follow up.

DETAILED DESCRIPTION:
Trauma is the leading cause of death worldwide in patients aged 1-45 years. Injuries and violence contribute to approximately 10% of all disability-adjusted life years globally. In Norway, approximately 10,000 patients are admitted to hospital annually due to trauma, with 66% being male. The mean age is 43 years for male and 48 years for female, indicating a relatively young patient population compared to other medical cohorts. The socioeconomic and functional implications of trauma are significant. With the expected demographic shift toward an aging population in Norway, the incidence of trauma among older adults is also expected to increase, placing greater demands on in-hospital trauma and rehabilitation services. Socioeconomic status, gender and age have been identified as key predictors of long-term outcomes following trauma, with female and individuals with lower education levels or ongoing compensation claims often reporting poorer outcomes.

While mortality rates are decreasing due to advancements in trauma systems, prevention strategies and medical care, a significant proportion of trauma survivors experience longterm disabilities, reduced quality of life, and difficulties in returning to work. These consequences impose substantial burdens on individuals, families, and society. Considering these issues, a shift in focus is needed-from survival alone to long-term functional recovery and quality of life after trauma.

Severe trauma often requires long-term follow-up, both physically and psychosocially. Traditional follow-up is often fragmented and not tailored to individual needs. Digital patient monitoring and tailored information have the potential to improve patient pathways, but knowledge about how these are experienced by patients, relatives, and healthcare professionals is limited.

This study aims to investigate how early rehabilitation and patient-centred care pathways can improve short and long-term outcomes for trauma patients. The objectives of the POSTRAUMA-trial is to assess the efficacy of a tailored patient information and patient managed outpatient digital follow-up (I-POD), as an adjunct to standard treatment according to the national guidelines in the National Trauma Plan (NTP) among adult trauma patients in Norway. The main research question is whether participants in the intervention group have less disability and improved health-related quality of life 6 months after the accident compared to the control group which receives standard treatment alone?

The latter part of the trial is a qualitative study which will follow the consolidated criteria for reporting qualitative studies (COREQ). SI will through in-dept and semi-structured interviews explore the participants experiences following trauma in general, and more specific to evaluate how the written patient information and digital follow-up was perceived. The SI will encourage the participants to talk about issues regarding this by asking open-ended questions in one-to-one interviews. The illness trajectory framework will be used as a theoretical framework, along with the WHOs International Classification of Functioning, Disability and Health (ICF) to ensure that preinjury, physical and biopsychosocial factors are evaluated.

ELIGIBILITY:
Inclusion Criteria:

* 16 years or older
* Fulfils the national criteria for TTA and admitted to HUS following trauma
* Included in NTR database
* Able to give informed consent

Exclusion Criteria:

* 15 years or younger
* Not included in NTR database
* Deceased before discharge from the hospital.
* Not able to give informed consent
* Insufficient command of the Norwegian language
* Foreign tourists or nationals
* Suicide attempt or serious self-inflicted trauma
* Serious psychiatric disorders or serious ongoing substance abuse

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 256 (Estimated)
Dates: Start 2026-03-02 (Estimated); Primary Completion 2027-03-02 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
EuroQol five-dimension utility score (EQ5D-index) from baseline to 6 months after the trauma in both groups. | From baseline to 6 months after the trauma
  The primary objective is to assess the efficacy of the I-POD-intervention as an adjunct to standard treatment after trauma according to national guidelines in adult patients in Norway. The efficacy is measured as the primary endpoint: EuroQol five-dimension utility score (EQ5D-index) from baseline to 6 months after the trauma in both groups. EQ5D-index ranges from - 0,59 (worst score) to 1 (perfect health, best score). 0 equals death. Baseline is defined as the time of inclusion.
  The I-POD intervention is a tailored patient Information and Patient-managed Outpatient Digital follow-up treatment.

SECONDARY OUTCOMES:
Differences in EuroQol five-dimension utility score (EQ5D-index) between the control group and the intervention group from baseline to 1 month and 12 months after the trauma. | Baseline to 1 month and 12 months after the trauma
  EQ5D-index ranges from - 0,59 (worst score) to 1 (perfect health, best score). 0 equals death.
Differences in HRQoL between the control group and the intervention group from baseline to 1 month, 6 months and 12 months after the trauma, measured by EuroQol visual analogue scale (EQ-VAS). | Baseline to 1 month, 6 months and 12 months after the trauma
  The EQ-VAS (EuroQol Visual Analogue Scale) is a standard tool used with the EQ-5D health questionnaire to measure a person's self-rated overall health on a vertical scale from 0 (worst imaginable health) to 100 (best imaginable health).
Differences in Return to work (RTW) between the control group and the intervention group at 1 month, 6 months and 12 months after the trauma by patient-reported data at 1 month, and 6 months and 12 months by NTR-data measured with dichotomous (yes/no) | Baseline to 1 month, 6 months and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Geir Arne Sunde, Ph.d, Principal Investigator — Haukeland University hospital, Surgical Department
Locations (1):
- Surgical Department, Haukeland University hospital, Bergen, Norway

IPD SHARING:
Plan to Share IPD: No
Sharing of privacy data is not within the scope of the ethical approval granted by REK West.